CLINICAL TRIAL: NCT07096388
Title: Evaluation Of Cost-Effectiveness Of Iliac Branch Endoprostheses: A Multi-Center, Retrospective-Prospective, Observational Study/ Eunet-Hta Core Model
Brief Title: Evaluation Of Cost-Effectiveness Of Iliac Branch Endoprostheses
Acronym: ECO-IBE
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Andrea Kahlberg (Other)
Responsible Party: Sponsor-Investigator, Prof. Andrea Kahlberg, Prof., IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: ECO-IBE STUDY
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Aorto-iliac Aneurysm
Keywords: endovascular repair; aorto-iliac aneurysm; iliac branch endoprotheses; open surgical repair
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular repair: Patients affected by an aorto-iliac aneurysm who received endovascular repair (with Iliac Branch Endoprosthesis)
  Interventions: Procedure: endovascular repair
- Open surgical repair: Patients affected by an aorto-iliac aneurysm who received an elective open surgical repair (aneurysmectomy and aortic reconstruction with a surgical graft)
  Interventions: Procedure: open surgical repair

INTERVENTIONS:
Procedure: endovascular repair — at first the iliac pathology main endovascular treatment was the graft stenting extended along the common and the external iliac artery with the embolisation of the internal iliac artery, with an high risk of pelvic ischemic complications, bowel ischemia, spinal cord ischemia, buttock claudication, erectile dysfunction. Nowadays, off-the-shelf endografts with a special design, the Iliac Branch Endoprosthesis, are available. These grafts, which preserve the hypogastric artery, avoiding complications due to its occlusion; they ensure better distal sealing by reducing the rate of type Ib endoleaks. The patient can be treated under local anesthesia and sedation or general anesthesia. Ultrasound-guided percutaneous access to one or both femoral arteries and, if needed, to the axillary or brachial artery is gained.
  Groups: Endovascular repair
Procedure: open surgical repair — in case of surgical repair of aorto-iliac aneurysms, general anesthesia is required. Access to the aorta can be achieved through a transperitoneal or retroperitoneal approach. A bifurcated graft is usually used for reconstruction as it is more similar to the native anatomical conformation, but it is not the only option. Although not mandatory, it may be necessary to revascularize one or both internal iliac arteries. This is a very complex surgical technique, challenging even for the most experienced operators due to the location of the iliac arteries. It is a procedure with a high risk of bleeding and mortality, and a high risk of damaging nearby structures such as the ureters and great veins. At the end of the procedure the patient is awake and is usually monitored in the recovery room and then translated to the ward, with fewer than 20% of patients needing Intensive Care Unit (ICU) admission.
  Groups: Open surgical repair

SUMMARY:
The study is a multi-center, voluntary observational study on an ambispective cohort of patients treated between January 2018 and December 2025.The study aims to enroll 300 patients (around 200 patients in the retrospective cohort and 100 patients in the prospective cohort). The study will include adult patients (≥ 18 years) of either sex submitted to open surgical repair or endovascular repair of an aorto-iliac aneurysm.The procedures and clinical evaluation included in this study correspond to current clinical practice. The assignment of the patient to a given diagnostic and/or therapeutic procedure is not linked to random allocation but is part of the ordinary therapeutic strategy provided for that patient; full freedom of choice as regards to the allocation of the patient to the diagnostic and therapeutic procedures is guaranteed for each case. Follow-up visits substantially correspond to current clinical practice or to the requirements of national and/or international guidelines. The administration of questionnaires, interviews, diaries, surveys of health economics and pharmacoeconomics, subjective assessments by the patient on their state of health, assessment scales and blood chemistry tests, the use of which is justified by the rationale of the study. The objectives of the study are the comparison of perioperative and late clinical success of repair procedure and comparison of cost-effectiveness of two precedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by an aorto-iliac aneurysm who received an elective open surgical repair (aneurysmectomy and aortic reconstruction with a surgical graft) or endovascular repair (with Iliac Branch Endoprosthesis)
* Adult patients ≥18 years
* Patients able to understand and sign the informed consent approved by the Ethics Committee of San Raffaele Hospital

Exclusion Criteria:

* Patients treated with a hybrid approach (concomitant open surgical and endovascular treatment)
* Patients treated with other endovascular techniques besides branched technology (e.g., physician-modified endografts, parallel grafts)
* Patients already submitted to prior open or endovascular repair for aorto-iliac aneurysm/prior aorto iliac aneurysm sac embolization
* Patients treated in urgent/emergent setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by an aorto-iliac aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of perioperative and late clinical success | 30 days 1 year 2 years
  Analysis of physiological parameters as Freedom from aorto-iliac related death, major adverse events (MAEs), and reintervention

SECONDARY OUTCOMES:
Comparison of cost-effectiveness | 30 days 1 year 2 years
  Measurements of structure, process and outcome relating to both direct and global costs (including major adverse events and reintervention-related costs)